CLINICAL TRIAL: NCT01964456
Title: "Narcisse & Echo : Self-consciousness and the Inter-subjective Body"
Brief Title: "Self-consciousness and the Inter-subjective Body"
Acronym: Narcisse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: The Volkswagen Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: D13-P001
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Anorexia Nervosa
Keywords: Bodily self-consciousness; intersubjective body; Anorexia Nervosa; Joint perception task; Interoceptive awareness
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients (Active Comparator): Patients suffering of anorexia
  Interventions: Other: Joint perception task; Behavioral: Body Shape Questionnaire; Other: Measure of the heart rate
- Control (Placebo Comparator): Subjects controls (not suffering of anorexia)
  Interventions: Other: Joint perception task; Behavioral: Body Shape Questionnaire; Other: Measure of the heart rate

INTERVENTIONS:
Other: Joint perception task
Behavioral: Body Shape Questionnaire
Other: Measure of the heart rate

SUMMARY:
The purpose of this study is to demonstrate that bodily self-consciousness is subjectively and inter-subjectively constituted and that some dimensions of the bodily self-consciousness are impaired in Anorexia nervosa.

DETAILED DESCRIPTION:
Anorexia nervosa is a severe psychiatric disorder, with high level of mortality. Anorexic patients often experience a serious disturbance in body and their own shape perception.

We hypothesize that bodily self-consciousness is co-constituted by four subjective dimensions which are all inter-subjectively open: in encountering others, one's body is experienced as

1. objectified,
2. the bearer of inter-subjective feelings,
3. an inter-subjective agent and
4. the anchor of an inter-subjectively negotiated perspective.

Across several experiments, we sought to determine which dimension of bodily self-consciousness is altered in Anorexia Nervosa compared to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Women
* From 18 to 35 years old
* Understanding and being fluent in French
* Hospitalized or followed in consultation for Anorexia nervosa (Restrictive Anorexia or Purge according to the MINI)
* Informed consent signed by the patient
* Diagnosis of Anorexia according to her psychiatrist (and confirmed by the DSM IV) with a BMI between 11 and 18.

Exclusion Criteria:

* Somatic Pathology (cancer, cardiac, renal or respiratory insufficiency, central neurological affection), evolutionary, or risking to be life-threatening within less than year
* Neurological Histories (neurological pathology susceptible to alter attentionnal capacities or field of vision and vision of colors (Encephalitis, Degenerative Brain tumour (méningiome, gliome, astrocytome), Congenital Neurodegenerative Pathology, Multiple sclerosis, Amyotrophic side Hardening, Epilepsy)
* Neuroleptic or psychotropic Treatment in doses inferring a slumber, a disorder of the concentration
* Dyschromatopsie
* No insurance
* Comorbidity of psychiatric type

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Joint perception task | 1 week
  Recording of the ocular behaviour in anorectic during the joint perception task.

SECONDARY OUTCOMES:
Body Shape Questionnaire | 1 week
  Body Shape Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mathias GOROG, MD, Principal Investigator — CHSA
Locations (1):
- Centre Hospitalier Sainte-Anne, Paris, France